CLINICAL TRIAL: NCT06528873
Title: NAZARÉ: Concurrent Optical and Magnetic Stimulation (COMS) for Treatment of Patients With Chronic Ulcers of Vascular Origin in a Real-world Setting Including Care at Patient's Home, a Prospective Randomized, Controlled, Assessor Blinded, Phase IV, Clinical Trial
Brief Title: COMS for Chronic Ulcers Treatment
Acronym: NAZARÉ
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Sebastian Probst (Other)
Collaborators: Medical University of Vienna (Other); University Hospital, Geneva (Other); Medical Centre Cité Générations (Unknown); Jura Hospital (Unknown); Clinique des Augustines (Unknown); Venenklinik Bellevue (Other); UniversitÃ¤tsklinikum Hamburg-Eppendorf (Unknown); Medical University of Graz (Other); UniversitÃ¤t Duisburg-Essen (Unknown); University Hospital, ZÃ¼rich (Unknown); Hospital Thun (Unknown)
Responsible Party: Sponsor-Investigator, Sebastian Probst, Professor of Tissue Viability and Wound Care, School of Health Sciences Geneva
Organization: School of Health Sciences Geneva (Other)
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Device Feasibility
Other Study IDs: NAZARÉ; PIOMIC (Other: PIOMIC)
Record Dates: First submitted 2024-07-26; First posted 2024-07-30 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Venous Leg Ulcer; Wound Heal; Magnetic Field Exposure
Keywords: Venous leg ulcer; optical stimulation; magnetic stimulation
MeSH Terms: conditions — Varicose Ulcer | interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: The COMS One therapy system is a CE-marked medical device for treating chronic leg and foot ulcers. It uses electromagnetic fields and photons non-invasively, non-ionizingly, non-thermally, and non-medicinally.
  The device transmits extremely low frequency (ELF) electromagnetic fields using a coil connected to a signal generator. It emits twenty trapezoid-shaped bursts per second, with the field's polarity switching every 2 minutes over a 16-minute session. The flux densities range from 0.4 mT to 1.6 mT in four-minute intervals.
  Photons are delivered via LEDs with peak wavelengths of 660 nm and 830 nm, targeting cytochrome C Oxidase. The light pulses at 1000 Hz, providing a radiant exposure of 2-5 J/cm² at a 1 cm distance from the skin.
  Technical details are in the IFU (100.0053_C_IfU).
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- usual care (No Intervention): Standard of Care treatment will be performed according to a provided standard of care manual according to most recent guidelines followed at each corresponding site (EWMA , S3-Leitlinie,…) and will proceed as follows:
  * Removal of old dressing
  * Application of analgesic if necessary
  * Debridement if necessary
  * Wound cleansing
  * Application of new dressing (according to the wound healing phases, medical prescription)
  * Application of compression therapy according to study standardized procedure (details in section 6.1).
  In the case the participant is at home, this procedure will be performed by a caregiver.
- COMS Therapy (Experimental): COMS treatment will be performed 2-3 times per week for at least 8 weeks, unless the wound heals sooner, with a minimum of 16 applications. Missed sessions can be made up in the 4-week follow-up period. Treatment will occur during standard care procedures, including dressing changes and debridement, and will follow these steps:
  Remove old dressing Apply analgesic if necessary Perform debridement if necessary Cleanse the wound Apply COMS One device Apply new dressing Apply compression therapy as per study procedures (section 6.1)
  If the patient is at home, a caregiver will perform this procedure. Study staff, including the PI, nurses, and caregivers, will receive training and a step-by-step document on using the COMS One device.
  Interventions: Combination Product: Concurrent optical and magnetic stimulation (COMS) treatment

INTERVENTIONS:
Combination Product: Concurrent optical and magnetic stimulation (COMS) treatment — COMS treatment will be performed 2-3 times per week for at least 8 weeks, unless the wound heals sooner, with a minimum of 16 applications. Missed sessions can be made up in the 4-week follow-up period. Treatment will occur during standard care procedures, including dressing changes and debridement, and will follow these steps:
  Remove old dressing Apply analgesic if necessary Perform debridement if necessary Cleanse the wound Apply COMS One device Apply new dressing Apply compression therapy as per study procedures (section 6.1)
  If the patient is at home, a caregiver will perform this procedure. Study staff, including the PI, nurses, and caregivers, will receive training and a step-by-step document on using the COMS One device.
  Arms: COMS Therapy

SUMMARY:
Chronic leg and foot ulcers are defined as wounds that fail to heal in a timely manner, typically persisting for over 4 to 8 weeks without substantial healing despite standard care. These ulcers often result from macro- and microvascular disorders, the most common being chronic venous insufficiency (CVI), alone or with peripheral artery disease (PAD) or microangiopathy. Despite different causes, chronic vascular-origin wounds share similar biological traits and require the same physiological processes for healing.

Vascular issues hinder blood perfusion, reducing oxygen, nutrients, and growth factors, leading to decreased energy metabolism and impaired cell functions necessary for proliferation, extracellular matrix production, angiogenesis, and tissue regeneration. Reduced blood supply also limits leukocyte function, compromising the immune response and leading to persistent inflammation and infection. Consequently, these wounds cannot effectively heal, showing prolonged inflammation, persistent infections, and cellular senescence.

Best practice wound care includes compression therapy and physical activity for venous ulcers, and angioplasty, surgery, or bypass for arterial ulcers. These treatments aim to improve blood flow, reduce venous stasis, and enhance venous return. Compression therapy and physical activity lower hydrostatic pressure in the lower limb, while angioplasty and surgery remove arterial blockages or create new blood flow routes.

Recent studies highlight the role of mechano-sensitive (MS) ion channels in skin cell processes and their dysfunction in dermatological disorders. Magnetic stimulation can activate MS TRCP1 channels, enhancing mitochondrial respiration and mitochondriogenesis via the Ca2+/CalModulin(CaM)/NFAT/PGC-1α pathway. Ca2+-activated calmodulin also catalyzes nitric oxide (NO), promoting vasodilation and tissue perfusion.

Bimodal red and near-infrared photobiomodulation can further increase mitochondrial respiration and ATP production by activating Cytochrome C oxidase and mitigating NO-induced downregulation. This synergistic mechanism of concurrent optical and magnetic stimulation (COMS) may amplify Ca2+ and NO-mediated processes like cell proliferation, migration, vasodilation, and angiogenesis while resolving inflammation. Thus, COMS may offer a promising therapy for chronic, inflammation-prone wounds.

The effectiveness of COMS has yet to be validated in large-scale studies. This proposal aims to assess the impact of COMS therapy combined with standard care versus standard care alone on healing, wound closure, recurrence, pain, quality of life, economic outcomes, and device usability in patients with venous leg ulcers (VLU) and VLU associated with PAD in a large-scale multicentric randomized controlled trial.

DETAILED DESCRIPTION:
Background: Chronic leg and foot ulcers are defined as wounds which fail to proceed through phases of wound healing in an orderly and timely manner to produce a durable structural functional and cosmetic closure. Depending on care setting / geographical region, wounds are considered chronic if they persist over more than 4 to 8 weeks with no substantial wound healing under standard of care (SOC) treatment regimen.

Among the most frequent causes for a delayed wound healing process are macro- and microvascular disorders. The most common is a chronic venous insufficiency (CVI), either as standalone or in combination with peripheral artery disease (PAD) or microangiopathy. Despite their differences in etiology, chronic wounds of vascular origin share similar biological features and require promotion of the same physiological processes for wound healing. The vascular constraints reduce blood perfusion and hinder appropriate cellular supply with oxygen, nutrients, and growth factors. This leads to decreased energy metabolism and therefore impaired cellular performance required for cell proliferation, extracellular matrix production, angiogenesis, and tissue regeneration. Additionally, reduced vascular supply decreases the number and ability of leukocytes to engage oxidative bursts, limiting the capacity for efficient pathogen destruction and leading to tissue devitalization. Consequently, the immune response becomes insufficient to deal with the local pathogen load, leading to ongoing inflammation in the wound area. In summary chronic wounds of vascular origins are unable to run through processes of wound healing, showing an inability to respond to local reparative stimuli of the wound environment, prolonged inflammation, persistent infections, and cellular senescence.

Best practice wound care emphasizes the utilization of compression therapy and physical activity for leg ulcers of venous etiology and angioplasty, surgery, or bypass operation for leg ulcers of arterial etiology, both axes of care being guided by the integration of healthcare professionals' clinical expertise with the best available clinical evidence. Compression therapy and physical activity facilitate wound healing by reducing hydrostatic pressure in the lower limb, mitigating venous stasis, and enhancing venous return. To improve the blood supply to the ulcer, angioplasty and surgery aims to clear out a blockage from a leg artery (endarterectomy), while bypass operation aims to put in a new route for blood flow in the leg.

Concurrent Optical and Magnetic Stimulation Recent publications have demonstrated the importance of mechano-sensitive (MS) ion channels in regulating processes such as skin cell proliferation, differentiation and barrier formation and linked their dysfunction to dermatological disorders. Magnetic stimulation has been shown to activate mechanosensitive TRCP1 channels, whereby the resulting ion channel-mediated calcium fluxes stimulate mitochondrial respiration and associated mitochondriogenesis through activation of the Ca2+/CalModulin(CaM) /NFAT/PGC-1α pathway. Ca2+-activated calmodulin has also been shown lead to the catalyzation of nitric oxide (NO), a potent mediator for vasodilation and tissue perfusion.

The concurrent bimodal red and near-infrared photo biomodulation, can further increase mitochondrial respiration and intracellular ATP production through activation of the Cytochrome C oxidase and mitigating its downregulation by increased levels of intracellular NO through its photo dissociation. Through this synergistic mechanism COMS may offer a therapeutic option for amplifying Ca2+ and NO mediated processes such as cell proliferation, migration, vasodilation, and angiogenesis while helping to shift the cytokine profile towards resolution of inflammation. Therefore, COMS may offer a promising therapeutic approach to enable the transition toward healing of therapy refractory wounds that tend to stay in inflammatory phase. The effectiveness of COMS has not yet been tested in a large-scale study. We propose here to assess the impact of COMS therapy+SOC versus SOC only, on healing, wound closure, wound recurrence, pain, quality of life, economic outcomes and device usability, in patients with venous leg ulcers (VLU) and VLU associated with PAD, in a large-scale multicentric randomized controlled trial.

Design: This study is a post market, phase IV clinical trial. A multicentric randomized controlled trial design will be used. 122 consecutive eligible patients with VLU or VLU associated with PAD, cared in outpatient or home settings in Switzerland (6 sites), France (1 site), Germany (2 sites) and Austria (2 sites), will be included and randomly allocated to one of the two study groups. Half of the participants will receive the standard of care (control group) and the other half will receive the standard of care, supplemented with COMS treatment during the 8 first week's post-inclusion (intervention group). Total study duration for each participant will be 24 weeks.

The intervention is single-blinded, i.e. it not blinded to participants and health care professionals but blinded to data assessors. Analysis:

The entire sample (intervention and control groups) will be described, according to the data level, in terms of their demographic and health data, using descriptive statistics. For the analysis of the different outcomes, the proportions or mean values will be compared between control and intervention groups by using classical tests of hypotheses. Additional analyses will be conducted to assess the change of the wound size over time and to compare groups. The statistical software for data science STATA 17.0 SAS version 9.4 or later (SAS Institute Inc., Cary, NC) will be used for data analysis.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed leg Ulcer of vascular origin (venous or mixed venous-arterial) without severe arterial insufficiency. Diagnosis of leg ulcer is based on angiological tests carried out at a given time, regardless of whether it is recent or older.
* Ulcer area between 2 - 50 cm2 after debridement
* Patients are older than 18 years of age.
* Chronic ulcer(s) with duration greater than 30 days and less than 2 years (continuous duration)
* If more than one ulcer is present, the target ulcer may be chosen based on the investigator's preference. However, the target ulcer must have a spatial distance of at least 5cm from all other ulcers so that measurements can be carried out accurately even in case an ulcer is growing in size.
* For diabetic patients: well-controlled diabetic mellitus (HbA1c ≤ 8%, historical results <3 months is acceptable)
* Adequate vascular perfusion as evidence by: ABI > 0.5 and < 1.30, ankle artery pressure >60 mmHg (historical results <3 months is acceptable).
* Women of childbearing age must agree to use adequate method of contraception
* Informed consent as documented by signature of the participant or a LAR, and being able to understand German or French language and follow the study protocol (cognition)

Exclusion Criteria:

* Women who are pregnant or breastfeeding (Women of childbearing potential need to perform a pregnancy test (urine test) within 24 hours prior to the study intervention and need at least one simple acceptable contraceptive method)
* Suspected skin cancer, or documented history of skin cancer or any other localized cancer, precancerous lesions or large moles in the areas to be treated.
* Use of photosensitizing agents or medications
* The patient is undergoing severe endogenous or drug immunosuppression
* Decompensated heart failure (NYHA III-IV)
* Patient with chronic renal insufficiency currently undergoing dialysis.
* Wounds with >30% wound area reduction in the last 2 weeks while receiving optimal standard of care (SOC) prior to randomization
* The patient is receiving systemic antibiotic treatment or is receiving/needing antibiotic wound therapy in/near the wound at inclusion
* The patient has received one of the following treatments in the last 2 weeks:

Arterial interventions such as angioplasty or vascular surgery. Venous Interventions including venous angioplasty, sclerotherapy, stenting, or endovenous thermal or non-thermal ablation.

* Cell and tissue based therapies such as punch & skin grafts in general, placental based allografts, autologous skin substitutes, cellular and acellular dermal matrix, platelet rich plasma and stem cell therapies
* Advanced wound care therapies such as shock wave, cold plasma, electric stimulation, ultrasound, negative pressure wound therapy, nanotechnologies, oxygen therapies
* Participants that were previously included in this clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Percent wound area reduction | 24 weeks
  Percent wound area reduction (PWAR) at week 12 will be measured from pictures of the wound taken with ImitoWound research application. PWAR is computed as (Wound area at baseline - Wound area at 12 weeks) / Wound area at baseline.
  The picture of the wound will be taken after dressing removal, wound debridement (if applicable) and wound cleansing. ImitoWound research App will be used in a smartphone as instructed in supplier's wound imaging and measurement guidelines. The camera of the smartphone will be positioned 20 to 30 cm away from and parallel to the wound. A calibration marker (quick response [QR] code) will be positioned next to and in the same plane of the wound, and a photograph will be taken after recognition of the QR code by the Imito App, automatic wound measurement will take place. Study nurses will receive concise training and document with step-by-step procedure for how to use Imito App.

IPD SHARING:
Plan to Share IPD: Yes
Raw data will be shared using Yareta (https://yareta.unige.ch/home) a Swiss research platform using the FAIR priniples
Supporting Information: Analytic Code
Time Frame: from 2027 until 2029
Access Criteria: all researchers
URL: https://yareta.unige.ch/home